CLINICAL TRIAL: NCT04379752
Title: Using Indirect Cold Atmospheric Pressure Plasma (Plasma Activate Liquid) for the Treatment of Hair Loss
Brief Title: Cold Plasma to Treat Hair Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Peter C. Friedman (Industry)
Responsible Party: Sponsor-Investigator, Dr. Peter C. Friedman, President, The Skin Center Dermatology Group
Organization: The Skin Center Dermatology Group (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200501
Record Dates: First submitted 2020-04-30; First posted 2020-05-07 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold-atmospeheric pressure plasma activated solution (Experimental): Treatment arm subjects receive the trial intervention
  Interventions: Device: Cold-atmospeheric pressure plasma activated aqueous-alcohol solution treatment

INTERVENTIONS:
Device: Cold-atmospeheric pressure plasma activated aqueous-alcohol solution treatment — Cold plasma is generated and applied to carrier liquid. Subjects are provided with the liquid to apply to the treated area

SUMMARY:
Self applied cold plasma activated medium used for androgenetic alopecia

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild-to moderate androgenetic alopecia
* ability of applying treatment regularly
* ability to keep in-person follow-up appointments

Exclusion Criteria:

* any inflammatory scalp condition
* starting or discontinuing any hair loss treatments within 6 months of start date
* allergy to any components of the carrier solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Presence of detectable hair growth | 3 months and 6 months
  Presence of hair growth is observed clinically. Evaluation may include photo comparison, hair count, trichoscopy

SECONDARY OUTCOMES:
Adverse effects related to the treatment | throughout study completeion, 6 months
  Patients are monitored for adverse effects, including but not limited to irritation, itch, inflammation, scaling, redness, rash, peeling, blistering

CONTACTS AND LOCATIONS:
Locations (1):
- The Skin Center Dermatology Group, New City, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan A, Malik S, Walia J, Fridman G, Fridman A, Friedman PC. Tolerability of Six Months Indirect Cold (Physical) Plasma Treatment of the Scalp for Hair Loss. J Drugs Dermatol. 2020 Dec 1;19(12):1177-1180. doi: 10.36849/JDD.2020.5186. PMID 33346510